CLINICAL TRIAL: NCT00190424
Title: Multicentric Randomized Phase 2. Immunotherapy With CpG-ODN in Malignant Glioblastoma
Brief Title: Randomized Phase 2 With CpG-ODN in Malignant Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P050305; ISOPS 3
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2005-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — CPG-oligonucleotide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- control (No Intervention)
- CpG-ODN (Experimental)
  Interventions: Drug: CpG-ODN

INTERVENTIONS:
Drug: CpG-ODN
  Arms: CpG-ODN

SUMMARY:
The purpose of this study is to determine whether the immunostimulating agent CpG-ODN is effective in the treatment of glioblastoma

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma
* Karnofsky Performance Status ≥ 60%

Exclusion Criteria:

* Severe or uncontrolled systemic disease
* Active auto-immune disease
* Uncontrolled epilepsia
* Platelets < 100 000/mm3 ; or Neutrophils <500 /mm3 ; or lymphocytes <300/ mm3

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2008-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Tolerance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre CARPENTIER, MD, PhD, Principal Investigator — Hopital Lariboisiere, Päris
Locations (2):
- France (2):
  - Hopital Salpetriere, Paris, Paris
  - Hopital Lariboisiere, Paris, Paris